CLINICAL TRIAL: NCT00602316
Title: Using Magnetic Resonance Techniques to Improve the Characterisation and Localisation of Breast Cancer. A Pilot Observational Study Testing the Accuracy of Multifunctional Magnetic Resonance Techniques in Predicting the Presence, Distribution and Nature of Breast Lesions in Women With Known Breast Cancer
Brief Title: Multifunctional Magnetic Resonance Imaging in Predicting Breast Lesions in Women Undergoing Mastectomy for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000581176; RMH-CCR2995
Record Dates: First submitted 2008-01-16; First posted 2008-01-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: gadolinium-chelate
Procedure: conventional surgery
Procedure: magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as multifunctional magnetic resonance imaging, may help doctors learn the extent of disease and plan the best treatment.

PURPOSE: This clinical trial is studying how well multifunctional magnetic resonance imaging works in predicting breast lesions in women undergoing mastectomy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the accuracy of multifunctional magnetic resonance (MR) in detecting, localizing, and characterizing satellite lesions in relation to an index breast tumor in order to improve definition of clinical target volume after local excision.

OUTLINE: Patients receive an injection of gadolinium chelate and undergo multifunctional magnetic resonance (MR) imaging, including dynamic contrast-enhanced MR, hydrogen-MR spectroscopy, and diffusion-weighted MRI, of the ipsilateral breast within 4 weeks before surgery. Patients undergo a mastectomy as planned. The resected specimen is photographed, and a histopathological analysis is performed consisting of the size and grade (if pre-invasive or invasive disease) of each satellite lesion, classification of benign satellite lesions, dimensions of each lesion, distance from the edge of the index tumor to the center of each satellite lesion, and the distance from the center of the surface of the nipple to the center of each lesion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-confirmed invasive ductal carcinoma of the breast
* Unifocal disease as defined by clinical examination, mammography, and ultrasound
* Patient must be proceeding to mastectomy
* Hormone receptor status unknown
* No T4d or multifocal disease (as defined on conventional imaging)
* Index tumor ≤ 4 cm in diameter

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Female
* No claustrophobia
* No cup size of DD or greater

PRIOR CONCURRENT THERAPY:

* No prior surgery to ipsilateral breast
* No prior neoadjuvant chemotherapy
* No prior ferromagnetic implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of magnetic resonance (MR) techniques in detecting histopathologically-identified multifocal and multicentric lesions

SECONDARY OUTCOMES:
Closeness of agreement between MR techniques and histopathology in localizing satellite lesions relative to the index tumor
Assessment of distribution of satellite lesions in relation to index tumor
Correlation between histopathological characteristics and signal changes on multifunctional MR

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kirby — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom